CLINICAL TRIAL: NCT03771027
Title: Evaluation of the Effectiveness of the Low FODMAP Diet in the Treatment of Functional Abdominal Pain in Children
Brief Title: Therapeutic Effect of the Low FODMAP Diet in Children With Functional Abdominal Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Katarzyna Boradyn, Principal Investigator, University of Warmia and Mazury
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/17/N/NZ5/02596
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Functional Abdominal Pain Syndrome
Keywords: low FODMAP diet; functional abdominal pain; children

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP diet group (Experimental): four weeks of the low FODMAP diet based on Monash University low FODMAP diet App.
  Interventions: Other: The low FODMAP diet.
- Control group (Active Comparator): four weeks of the diet based on NICE guidelines and contained products with different FODMAP content
  Interventions: Other: The diet based on NICE guidelines.

INTERVENTIONS:
Other: The low FODMAP diet. — The low FODMAP group had reduced the intake of FODMAP. Children received 3 main meals and 2 snacks daily prepared by the catering company according to the Human Nutrition Recommendations for Polish Population. The dietary intervention lasted four weeks.
  Arms: Low FODMAP diet group
Other: The diet based on NICE guidelines. — The control group based on NICE guidelines received diet contained products with different FODMAP content. Children received 3 main meals and 2 snacks daily prepared by the catering company according to the Human Nutrition Recommendations for Polish Population. The dietary intervention lasted four weeks.
  Arms: Control group

SUMMARY:
Diet components are important factors in pathogenesis of functional gastrointestinal disorders, especially in the irritable bowel syndrome. Fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAP) are a group of short chain, poorly absorbed and osmotically active carbohydrates, which can induce gastrointestinal symptoms because of rapid fermentation in different segments of the gut. Low FODMAP diet is a novel treatment option with proven efficacy in reducing symptoms of functional gastrointestinal disorders in adults. Conversely, although functional abdominal pain is a common health problem in children, the efficacy of a low FODMAP diet remains understudied in this population.

The aim of this study was to compare the effects of two diets: a low FODMAP diet and a diet based on standard dietary advice of the National Institute for Health and Care Excellence (NICE), on abdominal symptoms in children with functional abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

* functional abdominal pain according to Rome III criteria
* consent to participate in the study
* positive decision of gastroenterologist concerning enrolment of the patient to the trial

Exclusion Criteria:

* organic causes for gastrointestinal tract disorders,
* occurrence of an abdominal migraine, IBS, food allergies or intolerances, other significant disorders, acute infection
* antibiotic treatment within the last 8 weeks

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Assessment of abdominal pain severity | 6 weeks
  Wong-Baker FACES Pain Rating Scale where 0 = no hurt and 10 = hurts worst was used for assessed severity of abdominal pain during the 6-week study period (2 weeks before and 4 weeks during the diet)

SECONDARY OUTCOMES:
Assessment of abdominal pain and defecation frequency | 6 weeks
  Abdominal pain and defecation frequency were recorded as number per day.

OTHER OUTCOMES:
Assessment of stool consistency | 6 weeks
  Stool consistency was assessed using the validated Bristol Stool Form Scale. Type 1 or 2 were classified as the hard or lumpy stool, type 6 or 7 as the loose or waterly stool, and type 3-5 as the normal stool.
Assessment of nutritional status | 4 months
  Parameters of nutritional status before diet: weight (kilograms), height (meters).
Assessment of physical activity | 4 months
  The level of physical activity was established used the MVPA indicator (Moderate to Vigorous Physical Activity)
Assessment of well-being of the patient | 3 weeks
  Declarations of parents about symptoms changes in children during diet intervention based on a seven-point Likert scale (from 'much worse' to 'never occurred')

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna M Boradyn, MSc, Principal Investigator — Department of Human Nutrition, Faculty of Food Science, University of Warmia and Mazury; Elżbieta Jarocka-Cyrta, Ph.D, Principal Investigator — Department of Pediatrics, Gastroenterology and Nutrition, Collegium Medicum Faculty of Medicine, University of Warmia and Mazury; Katarzyna E Przybyłowicz, Ph.D, Principal Investigator — Department of Human Nutrition, Faculty of Food Science, University of Warmia and Mazury
Locations (2):
- Poland (2):
  - Regional Specialized Children's Hospital, Olsztyn
  - University of Warmia and Mazury, Olsztyn

IPD SHARING:
Plan to Share IPD: No